CLINICAL TRIAL: NCT00263614
Title: A Cross Sectional and Retrospective Evaluation in HBeAg-Positive or HBeAg-Negative Chronic Hepatitis B (CHB)Patients With Evidence of HBV Replication and Normal or Minimally Elevated Liver Transaminases(The MELT Study).
Brief Title: Evaluation of Chronic HBV Patients w/Evidence of HBV Replication and Normal or Minimally Elevated Liver Transaminases.
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Other Study IDs: GS-US-103-0143
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To determine whether HBeAg-positive and HBeAg-negative patients with HBV DNA greater than or less than 5 log10 and 4 log10 copies/mL, respectively, and with normal or minimally elevated liver transaminases have histological evidence of active liver disease.

DETAILED DESCRIPTION:
To determine whether HBeAg-positive and HBeAg-negative patients with HBV DNA greater than or less than 5 log10 and 4 log10 copies/mL, respectively, and with normal or minimally elevated liver transaminases have histological evidence of active liver disease.

ELIGIBILITY:
Inclusion Criteria: Patients must meet all of the following inclusion criteria to be included in this study:

Age greater than or equal to 18 years. Documented laboratory diagnosis of HBV infection (HBsAg positive) at least 6 months prior to inclusion in this study. Treatment naive, HBeAg-positive and HBeAg-negative patients. At least one liver biopsy specimen obtained in 2004 and/or 2005 (post diagnosis) that is available for evaluation by an independent pathologist. Gilead may allow enrollment of subjects with biopsies available from 2003. An adequate section of a biopsy for the purposes of this study should have at least 1 cm of the needle core of tissue on the slide. HBV DNA greater than or less than 5 log10 copies/mL for HBeAg-positive and greater than or less than 4 log10 copies/mL for HBeAg negative patients. A minimum of two normal or minimally elevated hepatic transminases (ALT) values that are at least 3 months apart during 2004 and/or 2005. Gilead may allow enrollment of subjects with values available from 2003. Minimally elevated ALT is defined as between lower limit of normal (LLN) and 1.2 times upper limit of normal (ULN) for HBeAg-positive and between lower limit of normal (LLN) and 1.5 times upper limit of normal (ULN) for HBeAg-negative patients. Child-Turcotte-Pugh score less than 7 and no evidence of ascites, variceal bleeding, or hepatic encephalopathy or impaired clotting function within 12 months prior to the Enrollment Visit.

Exclusion Criteria:Patients who meet any of the following criteria are excluded from the study:

History or evidence of HIV, hepatitic C, or hepatitis D. Other causes for liver disease other than hepatitis B, including but not limited to: hemochromatosis, Alpha-1 antitrypsin deficiency, Wilson's disease, Drug-related liver disease, Autoimmune hepatitis, Alcoholic liver disease, Obesity-induced liver disease (nonalcoholic seatohepatitis, NASH). History of, or current alcohol or substance abuse judged by the investigator to potentially interfere with laboratory or biopsy results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-12; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Flaherty, PharmD, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Inc., Foster City, California, United States

REFERENCES:
- [Derived] Hu KQ, Schiff ER, Kowdley KV, Min AD, Shiffman ML, Lee WM, Goodman ZD, Dau LO, Peschell KJ, Fagan EA, Flaherty JF. Histologic evidence of active liver injury in chronic hepatitis B patients with normal range or minimally elevated alanine aminotransferase levels. J Clin Gastroenterol. 2010 Aug;44(7):510-6. doi: 10.1097/MCG.0b013e3181d34c65. PMID 20179614
- See also: Gilead Sciences, Inc. website — http://www.gilead.com